CLINICAL TRIAL: NCT06827730
Title: PoCUS Impact on the Diagnostic Approach for Thoracic and Abdominal Pain in the ED
Acronym: DATAPUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: APHP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DATAPUS
Record Dates: First submitted 2025-01-24; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Pain; Thoracic Pain
Keywords: thoracic pain; abdominal pain; point of care ultrasound; diagnostic approach
MeSH Terms: conditions — Abdominal Pain; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with thoracic or abdominal pain (Other): Patients presenting at the emergency department complaining of non-traumatic thoracic or abdominal pain for less than 72 hours and for whom no previous complementary examinations were performed to investigate the pain.
  Interventions: Diagnostic Test: Point of care ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound — The investigator uses PoCUS to investigate thoracic or abdominal pain after anamnesis and clinical examination. The investigator reports the anamnesis, clinical examination, and PoCUS results in the patient's medical file. PoCUS images are recorded according to the procedures of the study centers and the capacities of the ultrasound machines.
  Other Names: PoCUS

SUMMARY:
Many medical specialties and paramedical fields are increasingly using point-of-care ultrasound (PoCUS). In daily practice, thoracic and abdominal pain constitute a significant portion of emergency department consultations. PoCUS can be employed in various ways during thoracic and abdominal physical examinations. Most scientific societies advocate for its use to address specific clinical questions rather than to provide a definitive diagnosis.

The integration of PoCUS into clinical examinations raises the question of its effectiveness in improving the diagnostic approach, rather than its diagnostic accuracy alone. Given the broad spectrum of differential diagnoses for thoracic and abdominal pain, this multicenter prospective study protocol aims to evaluate how PoCUS enhances the diagnostic approach for patients presenting with these symptoms in the emergency department.

To assess the contribution of PoCUS, three members of an adjudication committee will blindly choose between two case report forms reporting the planned diagnostic approach for each patient: one completed before PoCUS and the other after its use by the investigator handling the case. The hypothesis that PoCUS improves the diagnostic approach by 60% will be reached if 60% of the improved diagnostic approaches favor the case report form filled out after PoCUS.

DETAILED DESCRIPTION:
1. Background

   Point-of-care ultrasound (PoCUS) is increasingly utilized across various medical and paramedical fields. As a fundamental component of clinical evaluation alongside inspection, palpation, percussion, and auscultation, PoCUS has become indispensable in daily clinical practice enhancing differential diagnosis. In a position statement published in 2015, the American Academy of Emergency Medicine followed by the European Federation of Societies for Ultrasound in Medicine and Biology in 2016 recommended the inclusion of PoCUS in the curricula of medical schools to improve core concepts learning and enhance students' understanding of physical examinations. The integration of PoCUS into clinical practice emphasizes its role in refining the diagnostic approach rather than merely focusing on its diagnostic accuracy.

   In daily practice, thoracic pain accounts for about 5% and abdominal pain for 7% to 10% of emergency department consultations. PoCUS can be used in many ways during thoraco-abdominal physical examinations, and most scientific societies encourage its use to address a specific clinical question rather than to provide a diagnosis. For this reason, it is important to focus on the impact of PoCUS on the overall diagnostic approach rather than solely on its diagnostic accuracy. The diagnostic approach includes selecting diagnoses for differential diagnosis, choosing appropriate treatments, and determining necessary complementary examinations, all conducted following the clinical examination.

   The primary objective of this study is to evaluate the contribution of PoCUS to the diagnostic approach of patients presenting to the emergency department with thoracic or abdominal pain. Secondary outcomes include the influence of PoCUS on the selection and number of diagnoses in the differential diagnosis, the number of additional treatments or complementary diagnostic examinations, its impact on physicians' confidence in their diagnostic approach, the influence of patient characteristics or PoCUS findings on the primary outcome and evaluate financial aspects.
2. Method

   • This study is an interventional multicenter international prospective study evaluating the contribution of PoCUS on the diagnostic approach for patients presenting at the emergency department with thoracic or abdominal pain.

   The interventional aspect of the study is secondary to the one-month follow-up of patients based on patients' medical files and phone consultation to establish the final diagnosis. However, PoCUS is considered standard of care, as supported by clear guidelines that advocate for its integration into standard medical practice in both Europe and North America.

   Thoracic or Abdominal PoCUS will be performed according to an established protocol

   Prior to the study launch, all investigators will participate in a 2-hour refresher course on point-of-care ultrasound (PoCUS) of the thorax and abdomen. Each investigator is already familiar with PoCUS and uses it daily in their clinical practice. Investigators are required to hold a certification or a diploma in PoCUS. They will all be required to rate their comfort level with PoCUS on a Likert scale from 0 to 5, in response to the questions: "On a scale from 0 to 5, how comfortable are you with using PoCUS to evaluate the thorax?" and "On a scale from 0 to 5, how comfortable are you with using PoCUS to evaluate the abdomen?". The investigator will be selected if the comfort level is at 4 or 5.

   Patient eligibility will be determined by nurses at triage.

   Any patient presenting with thoracic or abdominal pain will be evaluated according to the following three questions:
   * Can you show me with your hand where is the pain located?
   * Have you been in pain for less than 72 hours?
   * Did you undergo any complementary medical examinations to evaluate the pain before coming to our emergency department? If the patient localizes the pain in the anterior thorax or the abdomen, has experienced pain for less than 72 hours, and did not undergo any complementary medical examinations, the triage nurse will call the study investigator. The triage nurse will then continue the triage process with no interference from the study investigator, give painkillers if required, and orientate the patient to the appropriate emergency department sector for medical consultation.

   Inclusion process Without interfering with the patient triage, the study investigator will assess the patient's eligibility, explain the study, and obtain a signed informed consent. The investigator will then verify the inclusion, non-inclusion and exclusion criteria and initiate the study process by taking charge of the patient and performing an anamnesis and clinical examination.

   The investigator will fill in the first part of the computerized CRF. After validation, no changes can be made by the investigator.

   Intervention process The investigator uses PoCUS. The investigator will fill in the second part of the computerized CRF. After validation, no changes can be made by the investigator.

   The investigator will then complete the third part of the computerized CRF comprising the PoCUS results.

   The investigator is not required to limit the PoCUS examination to the PoCUS protocol if the patient's care requires further PoCUS examinations. However, the rest of the PoCUS examination will be performed after the three sections of the CRF are completed and sealed.

   The investigator reports the anamnesis, clinical examination, and PoCUS results in the patient's medical file.

   PoCUS images are recorded according to the procedures of the study centers and the capacities of the ultrasound machines.

   Evaluation process The first adjudication committee (2 members) will determine the final diagnosis based on the patient's medical records and a follow-up phone consultation conducted at 1-month follow-up. They have no access to the study data except for question relating to the 1-month follow-up.

   After validating the final diagnosis and anonymizing the data, the second adjudication committee (3 members) will independently evaluate the diagnostic approaches. This second adjudication committee is blind to the intervention but aware of final diagnosis. Before assessing the diagnostic approaches, CRFs are anonymized and randomly ordered using the "Randomizer for Clinical Trial Lite" Medsharing, Fontenay-Sous-Bois, France. For each included patient, only the study coordinator is aware of the order of the diagnoses approaches (one before and one after PoCUS). The members of the adjudication committee are therefore not aware of which diagnostic approach is before or which is after PoCUS.

   After assessing the two diagnostic approaches, two members of the second adjudication committee will determine which diagnostic approach is superior or if the two approaches are equivalent. The third member oversees the adjudication in case of discrepancies.

   Study members
   * Patients Patient eligibility as well as the inclusion, non-inclusion and exclusion criteria are reported above. During the entire study, patients have the right to stop participating.
   * Triage nurses Triage nurses notify the investigator from the triage section of the emergency department. They do not play a specific role in the study inclusion process. The study inclusion process cannot interfere with the triage.
   * Investigators The investigators are all emergency physicians who are familiar with PoCUS of the thorax or of the abdomen and who underwent a 2-hour refresher course on the PoCUS process used for this particular study.
   * Adjudication committee members

     * Adjudication committee 1 Two emergency physicians confirm the final diagnoses of patients according to their medical file and a phone consultation at 1-month follow-up. The two physicians work together to determine the correct final diagnosis that explains the pain that led to the emergency department consultation. A third member may be required to adjudicate any discrepancies.
     * Adjudication committee 2 Two emergency physicians who are blind to the study intervention independently choose the better diagnostic approach according to final diagnosis and a third one adjudicate in case of discrepancy. If no diagnostic approach is considered better, the diagnostic approaches are considered equivalent.

   The diagnostic approach will be considered superior if the differential diagnosis, treatment choices and complementary investigations planned are deemed more accurate considering the final diagnosis.

   • Research associate Research associates will oversee the 1-month follow-up of patients and will help with the study coordination and launch at the different study centers.

   • Biostatisticians Through the "Support en Methodologie et Calculs Statistiques" of the Université Catholique de Louvain, a biostatistician will perform the statistical analyses of this study.

   f. Sample size

   A total of 369 (323) patients are needed to show a 60% (70%) improvement in the diagnostic approach with a power of 0.8 and an alpha value of 0.05. Considering an attrition rate of 10%, the sample size needed to perform this study is 406 (356) patients. An 60% improvement in the diagnostic approach is based on previous publications showing a 45% to 82% rate of diagnostic improvement after PoCUS use in non-traumatic abdominal pain.

   g. Statistical method

   The software IBM SPSS statistics 26.0 (SPSS Inc., Chicago, IL, USA) will be used to analyze the data. Continuous variables describing the study population will be detailed using medians, standard deviations, and minimum and maximum values. Discrete variables will be reported by category as numbers and percentages. The χ² test of independence will be used for comparison between discrete variables. The Wilcoxon-Mann-Whitney test will be used for comparison between continuous variables. The significance level corresponds to a p-value of 0.05 or less. The 95% confidence intervals will be calculated using the mid-p exact value.

   Primary endpoint

   • Assessing the improvement of the diagnostic approach using PoCUS as part of the clinical examination for patients presenting at the emergency department with thoracic or abdominal pain

   o This will be evaluated using a proportion test performed according to the expected percentage of improvement (60%).

   Secondary endpoints
   * PoCUS influence on the number of diagnoses in the differential diagnosis, on the number of treatments and on the number of complementary examination(s)

     o Comparison of means, paired t-test if parametric data distribution, and Wilcoxon test for non-parametric data distribution
   * PoCUS influence on the physicians' coefficient of certainty regarding the diagnostic approach

     o χ² test
   * PoCUS influence on the physicians' coefficient of certainty regarding the final diagnosis if this diagnosis is part of the differential diagnosis established bedside

     o χ² test
   * PoCUS usefulness evaluated by the physician in charge (not useful, useful, very useful)

     o χ² test
   * Influence of PoCUS findings on the primary outcome (Positive PoCUS or negative PoCUS)

     o Proportion test
   * Influence of patients' characteristics (BMI, echogenicity, triage score, pain scale, final diagnosis) on the primary outcome

     * Proportion test
     * χ² test to evaluate the categories established in the subgroups compared to each other
   * Influence of PoCUS on financial aspects

     * Proportion test
     * χ² test to evaluate the categories established in the subgroups compared to each other
3. Data management

   1. Data collection

      All the data relating to this study will be collected on computerized CRF on REDcap (Research Electronic Data Capture) by the study investigator. Collected data will concern the clinical situation, patient characteristics, test results, and diagnostic approach associated with the coefficients of certainty of the physicians in charge as well as any questions relating to the bedside PoCUS. Any missing data will be collected from the medical file by the inclusion center's principal investigator, coordinating investigator, or research associates. The first adjudication committee will have access to the patients' anonymized medical files at 1-month follow-up to determine the final diagnoses. This committee will nevertheless not have access to the data collection dedicated to the study. This committee will process to confirmation of final diagnosis in the dedicated center. Files will be printed and anonymized previously to the committee evaluation.

      Patients will initially be identified on the CRF by their last name, first name, date of birth, file number from the institution where they were included, and an identification number of the study. This identification number will be comprised of a reference for the inclusion center and participant number. After the principal investigators or research associates complete the collection of missing data, patients will henceforth only be identified by their study identification number to anonymize the data.
   2. Data access

      A list of correspondence between the study identification number and the other identifying data will be kept under the responsibility of the project promoter. This list is kept for the statutory period of time provided for this type of research. The protection of the patients' personal data will be guaranteed by the European General Data Protection Regulation of 27 April 2016 (in application since 25 May 2018), the Belgian Law of 30 July 2018 on privacy protection with regard to the processing of personal data, and the Belgian Law of 22 August 2002 on patient rights.

      A certified good clinical practice will be used with a compliant electronic data management system. The system is connected to the clinical center database management system and protected by the personal identification of authorized users. This distinguishes between users and guarantees data safety.

      Any individual with direct access to the data shall take all the necessary precautions to ensure the confidentiality of the information relating to participants included in the study, particularly with regard to their identity and results. Any individual with direct access to data are subject to professional secrecy. They undertake to never divulge confidential information relating to the study participants and to guarantee the anonymization of the data before transferring it to the database manager and biostatistician. Any data disclosure required by the law or applicable regulations will be done if necessary.
   3. Data storage

   After completing the data collection and anonymizing the data, they will be added to a file (SPSS 26.0) with access limited by a password. This document will be owned by the project promoter represented by the study coordinator. This person ensures that the documents and data relating to the research are kept for 20 years in accordance with the applicable regulations. Coordinating investigators are responsible for keeping the essential study documents at the research site. If they leave the institution, they will delegate this responsibility to the project promoter in writing.
4. Ethics

Written documentation explaining the PoCUS procedure and the risks/benefits of undergoing PoCUS will be given to all participants. They will also receive an explanation about data protection.

Ultrasound technology does not put participants at risk during abdominal ultrasound. Indeed, physicians are required to observe the ALARA (as low as reasonably achievable) principle during clinical examinations. Signed written consent to participate in this study will be collected for each participant in Belgium and in France as recommended by the Additional Protocol to the Convention on Human Rights and Biomedicine Concerning Biomedical Research as well as by the Council of Europe's Steering Committee on Bioethics.

A study file including this protocol, a summary, and the CRF will be submitted to the ethics committees of each participating center. The research protocol will only begin if a favorable opinion is issued by the local ethics committees and by the ethics committee of the main center. Any substantial changes to the study file must be approved by the study promoter. Before any changes take place, all the ethics committees will need to give their approval. The project promoter will communicate the end date of the study to the ethics committees within a delay of 90 days. This date will correspond to the date of the last inclusion or, if appropriate, to the theoretical end date of the study in this protocol. If the inclusion number is not reached within 1 year, an extension request will be added to this protocol.

1. Compensation There is no compensation for the participants of this study.
2. Adverse event

   An adverse event is any untoward medical occurrence including the exacerbation of an existing condition that is not necessarily related to the study itself. Any incidental findings using PoCUS will be reported, and information will be given under medical confidentiality. The family physician will also be notified by telephone and by a consultation letter from the emergency department. All the results will be recorded confidentially in the patient's medical file. The reasons for losing participants to follow-up will also be mentioned.

   This is a clinical study. Right upper quadrant PoCUS is a non-invasive procedure for which no reported risk was identified in the current literature. In this study, patient management will always take priority over performing PoCUS.
3. Insurance Regarding the law of 7 May 2004, the project promoter will take out insurance to cover any risk incurred by the study's participants in Belgium. Another insurance will be taken by the different participating centers.

ELIGIBILITY:
Inclusion Criteria:

* > 17 years
* Thoracic or abdominal pain for less than 72 hours
* Signed informed consent

Exclusion Criteria:

* Reasons making abdominal ultrasound impossible
* Discovery of a pregnancy during emergency care
* Follow-up impossible at one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of superior diagnostic approaches post-PoCUS. | From enrollment to the completion of the one-month follow-up
  Percentage of superior diagnostic approaches post-PoCUS.
  For each patient included in the final analysis and based on the final diagnosis determined at the 1-month follow-up, three independent members of an adjudication committee will evaluate the two diagnostic approaches (pre-PoCUS and post-PoCUS) recorded in the case report forms (CRFs). The adjudication committee members will remain blinded to the intervention, ensuring they are unaware of whether the diagnostic approach occurred before or after PoCUS. For each patient, the committee, knowing the final diagnosis, will assess and determine which diagnostic approach is superior or if the two approaches are equivalent.

SECONDARY OUTCOMES:
PoCUS influence on the number of diagnoses in the differential diagnosis, on the number of treatments and on the number of complementary examination(s) | From enrollment to the completion of the one-month follow-up
  Absolute number before and after PoCUS
PoCUS influence on the physicians' coefficient of certainty regarding the diagnostic approach | From enrollment to the completion of the one-month follow-up
  Evaluation of % of certainty coefficient before and after PoCUS
PoCUS influence on the physicians' coefficient of certainty regarding the final diagnosis if this diagnosis is part of the differential diagnosis established bedside | From enrollment to the completion of the one-month follow-up
  Evaluation of % of certainty coefficient before and after PoCUS
PoCUS usefulness evaluated by the physician in charge | From enrollment to the completion of the one-month follow-up
  Number of PoCUS considered not useful, useful, very useful
Influence of PoCUS findings on the primary outcome (Positive PoCUS or negative PoCUS) | From enrollment to the completion of the one-month follow-up
  Influence of a positive or a negative PoCUS finding on the primary outcome
Impact of the body mass index level on the primary outcome | From enrollment to the completion of the one-month follow-up
  Subgroup analysis
Influence of PoCUS on financial aspects | From enrollment to the completion of the one-month follow-up
  Difference of costs of the diagnostic approach before and after PoCUS

CONTACTS AND LOCATIONS:
Overall Officials: Florence MV Dupriez, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ma IWY, Arishenkoff S, Wiseman J, Desy J, Ailon J, Martin L, Otremba M, Halman S, Willemot P, Blouw M; Canadian Internal Medicine Ultrasound (CIMUS) Group*. Internal Medicine Point-of-Care Ultrasound Curriculum: Consensus Recommendations from the Canadian Internal Medicine Ultrasound (CIMUS) Group. J Gen Intern Med. 2017 Sep;32(9):1052-1057. doi: 10.1007/s11606-017-4071-5. Epub 2017 May 11. PMID 28497416
- [Background] Cervellin G, Mora R, Ticinesi A, Meschi T, Comelli I, Catena F, Lippi G. Epidemiology and outcomes of acute abdominal pain in a large urban Emergency Department: retrospective analysis of 5,340 cases. Ann Transl Med. 2016 Oct;4(19):362. doi: 10.21037/atm.2016.09.10. PMID 27826565
- [Background] Kohn MA, Kwan E, Gupta M, Tabas JA. Prevalence of acute myocardial infarction and other serious diagnoses in patients presenting to an urban emergency department with chest pain. J Emerg Med. 2005 Nov;29(4):383-90. doi: 10.1016/j.jemermed.2005.04.010. PMID 16243193
- [Background] Atkinson P, Bowra J, Lambert M, Lamprecht H, Noble V, Jarman B. International Federation for Emergency Medicine point of care ultrasound curriculum. CJEM. 2015 Mar;17(2):161-70. doi: 10.1017/cem.2015.8. PMID 26052968
- [Background] Prosch H, Radzina M, Dietrich CF, Nielsen MB, Baumann S, Ewertsen C, Jenssen C, Kabaalioglu A, Kosiak W, Kratzer W, Lim A, Popescu A, Mitkov V, Schiavone C, Wohlin M, Wustner M, Cantisani V. Ultrasound Curricula of Student Education in Europe: Summary of the Experience. Ultrasound Int Open. 2020 Jun;6(1):E25-E33. doi: 10.1055/a-1183-3009. Epub 2020 Aug 31. PMID 32885138
- [Background] Nicholas E, Ly AA, Prince AM, Klawitter PF, Gaskin K, Prince LA. The Current Status of Ultrasound Education in United States Medical Schools. J Ultrasound Med. 2021 Nov;40(11):2459-2465. doi: 10.1002/jum.15633. Epub 2021 Jan 15. PMID 33448471
- [Background] Cantisani V, Dietrich CF, Badea R, Dudea S, Prosch H, Cerezo E, Nuernberg D, Serra AL, Sidhu PS, Radzina M, Piscaglia F, Bachmann Nielsen M, Ewertsen C, Saftoiu A, Calliada F, Gilja OH. EFSUMB Statement on Medical Student Education in Ultrasound [long version]. Ultrasound Int Open. 2016 Mar;2(1):E2-7. doi: 10.1055/s-0035-1569413. PMID 27689163
- [Background] Soucy ZP, Mills LD. American Academy of Emergency Medicine Position Statement: Ultrasound Should Be Integrated into Undergraduate Medical Education Curriculum. J Emerg Med. 2015 Jul;49(1):89-90. doi: 10.1016/j.jemermed.2014.12.092. Epub 2015 Apr 29. No abstract available. PMID 25934381
- [Background] Hayward SA, Janssen J. Use of thoracic ultrasound by physiotherapists: a scoping review of the literature. Physiotherapy. 2018 Dec;104(4):367-375. doi: 10.1016/j.physio.2018.01.001. Epub 2018 Feb 2. PMID 29958691
- [Background] Meadley B, Olaussen A, Delorenzo A, Roder N, Martin C, St Clair T, Burns A, Stam E, Williams B. Educational standards for training paramedics in ultrasound: a scoping review. BMC Emerg Med. 2017 Jun 17;17(1):18. doi: 10.1186/s12873-017-0131-8. PMID 28623905
- [Background] Dupriez F, Niset A, Couvreur C, Marissiaux L, Gendebien F, Peyskens L, Germeau B, Fasseaux A, Rodrigues de Castro B, Penaloza A, Vanpee D, Bobbia X. Evaluation of point-of-care ultrasound use in the diagnostic approach for right upper quadrant abdominal pain management in the emergency department: a prospective study. Intern Emerg Med. 2024 Apr;19(3):803-811. doi: 10.1007/s11739-023-03480-9. Epub 2023 Dec 2. PMID 38041765
- [Background] Jang T, Chauhan V, Cundiff C, Kaji AH. Assessment of emergency physician-performed ultrasound in evaluating nonspecific abdominal pain. Am J Emerg Med. 2014 May;32(5):457-60. doi: 10.1016/j.ajem.2014.01.004. Epub 2014 Jan 16. PMID 24529645